CLINICAL TRIAL: NCT06906783
Title: Comparison of Transtibial Pull Out Method And Suture Anchor Method in Surgical Treatment of Meniscus Extrusion
Brief Title: Transtibial Pull Out Method Versus Suture Anchor Method for Meniscus Extrusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammet Celik, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATAUNIORTHO
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Meniscal Extrusion; Meniscus Injury
Keywords: Meniscus Extrusion; Surgical Treatment; Transtibial Pull Out; Suture Anchor Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transtibial Pull Out Method (Active Comparator)
  Interventions: Procedure: Transtibial Pull Out Method
- Suture Anchor Method (Active Comparator)
  Interventions: Procedure: Suture Anchor Method

INTERVENTIONS:
Procedure: Transtibial Pull Out Method — The Transtibial Pull-Out Repair is a surgical technique used to fix posterior root tears of the meniscus, particularly in the medial meniscus. This method restores the hoop stress mechanism of the meniscus, which is essential for knee stability and function.
  Arms: Transtibial Pull Out Method
Procedure: Suture Anchor Method — The Suture Anchor Technique is an alternative to the Transtibial Pull-Out Method for repairing posterior meniscal root tears, especially in the medial meniscus. Instead of using a tibial tunnel, this technique fixes the meniscal root directly to the native footprint using suture anchors.
  Arms: Suture Anchor Method

SUMMARY:
The concept of meniscal extrusion has recently been recognized as an important pathological condition associated with meniscal dysfunction. Meniscal extrusion is the medial or lateral displacement of the meniscus beyond the edges of the tibial plateau. Some meniscal extrusions are physiologic, but large degrees of extrusion are thought to be pathologic.

Meniscal extrusion can vary in extent from minimal physiological extrusion to extrusions exceeding 10 mm. The generally accepted threshold value is considered to be 3 mm.

To date, the gold standard for measuring meniscal extrusion is T2-weighted MRI. MRI is valuable not only due to its ability to define other meniscal or knee pathologies but also because it provides good sensitivity and specificity.

Surgical treatment of meniscal extrusion is preferred in young, active, symptomatic patients and individuals with acute injuries. The treatment approach may vary depending on the underlying cause. One of these methods is centralization surgery, which aims to achieve the anatomical reduction of the extruded meniscus.

The aim of this study is to compare the functional outcomes of transtibial pull-out and suture anchor techniques used in centralization surgery and to contribute to standardization.

ELIGIBILITY:
Inclusion Criteria:

* Presence of meniscal extrusion greater than 3 mm on MRI scans
* Symptomatic complaints in the knee with extrusion

Exclusion Criteria:

* Malalignment greater than 5 degrees
* Presence of Kellgren-Lawrence grade 3-4 osteoarthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in the amount of meniscus extrusion in MR images. | From enrollment to the end of treatment at 12 months
  determine the change in the amount of meniscus extrusion in preoperative and postoperative 12th month MR images.

SECONDARY OUTCOMES:
Lysholm score | From enrollment to the end of treatment at 3, 6 and 12 months.
  The Lysholm score is a 100-point scoring system for examining a patient's knee-specific symptoms including mechanical locking, instability, pain, swelling, stair climbing, and squatting.
Tegner activity score | From enrollment to the end of treatment at 3, 6 and 12 months.
  The scale is numbered on a "0-10" format, with 10 being international soccer, and one being a person who is disabled from knee issues.
International Knee Documentation Committee (IKDC) Score | From enrollment to the end of treatment at 3, 6 and 12 months.
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet E Paksoy, Assoc.Prof., Study Director — Ataturk University
Locations (1):
- Ataturk University Hospital, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yan X, Sahu S, Li H, Zhou W, Xiong T, Chen S, Li C, Hao L. Arthroscopic meniscal posterior root repair combined with centralization reduces medial meniscus extrusion associated with posterior root tears: One-year clinical outcomes. Knee Surg Sports Traumatol Arthrosc. 2025 Aug;33(8):2825-2832. doi: 10.1002/ksa.12533. Epub 2024 Nov 14. PMID 39543774
- [Result] Zhou Y, Yang Q, Kang J, Xu J, Chen M, Wu C. Clinical effect of medial meniscus posterior root repair combined with centralization technique in the treatment of medial meniscus posterior root tears. BMC Musculoskelet Disord. 2024 Nov 30;25(1):982. doi: 10.1186/s12891-024-08125-2. PMID 39616323